CLINICAL TRIAL: NCT01064401
Title: Multicenter, Double-blind, Randomized, Parallel-group, Monotherapy, Active-control Study to Determine the Efficacy and Safety of Daclizumab High Yield Process (DAC HYP) Versus Avonex® (Interferon β 1a) in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Efficacy and Safety of BIIB019 (Daclizumab High Yield Process) Versus Interferon β 1a in Participants With Relapsing-Remitting Multiple Sclerosis
Acronym: (DECIDE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205MS301; 2009-012500-11
Record Dates: First submitted 2010-01-26; First posted 2010-02-08 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — daclizumab HYP; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daclizumab High Yield Process 150 mg SC (Experimental): Daclizumab High Yield Process (DAC HYP) 150mg subcutaneous (SC) injection once every 4 weeks plus placebo to IFN β-1a intramuscular (IM) injection once weekly for 96 to 144 weeks
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process); Drug: Interferon beta-1a Placebo
- IFN β-1a 30 µg IM (Active Comparator): Interferon beta-1a (IFN β-1a) 30 µg IM once weekly plus placebo to DAC HYP SC once every 4 weeks for 96 to 144 weeks
  Interventions: Biological: Interferon beta-1a; Drug: Daclizumab High Yield Process Placebo

INTERVENTIONS:
Biological: BIIB019 (Daclizumab High Yield Process) — Daclizumab High Yield Process for subcutaneous injection
  Other Names: DAC HYP
  Arms: Daclizumab High Yield Process 150 mg SC
Drug: Interferon beta-1a Placebo — Placebo to interferon beta-1a intramuscular injection
  Arms: Daclizumab High Yield Process 150 mg SC
Biological: Interferon beta-1a — Interferon beta-1a for intramuscular injection
  Other Names: Avonex; IFN β-1a
  Arms: IFN β-1a 30 µg IM
Drug: Daclizumab High Yield Process Placebo — Placebo to Daclizumab High Yield Process subcutaneous injection
  Arms: IFN β-1a 30 µg IM

SUMMARY:
The primary study objective is to test the superiority of Daclizumab High Yield Process (DAC HYP) compared to interferon β 1a (IFN β-1a) in preventing multiple sclerosis (MS) relapse in participants with relapsing remitting multiple sclerosis.

The secondary study objectives are to test the superiority of DAC HYP compared to IFN β-1a in slowing functional decline and disability progression and maintaining quality of life in this participant population.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS), and a cranial magnetic resonance imaging (MRI) demonstrating lesion(s) consistent with MS
* Must have a baseline Expanded Disability Status Scale (EDSS) between 0.0 and 5.0, inclusive
* Male subjects and female subjects of childbearing potential must be willing to practice effective contraception during the study and be willing and able to continue contraception for 4 months after their last dose of study treatment

Key Exclusion Criteria:

* Known intolerance, contraindication to, or history of non-compliance with Avonex® 30 µg
* History of treatment with Daclizumab High Yield Process (Dac HYP)
* History of malignancy
* History of severe allergic or anaphylactic reactions
* Known hypersensitivity to study drugs or their excipients
* History of abnormal laboratory results indicative of any significant disease
* History of human immunodeficiency virus (HIV) or other immunodeficient conditions
* History of drug or alcohol abuse (as defined by the Investigator) within the 2 years prior to randomization
* History of seizure disorder or unexplained blackouts OR history of a seizure within 6 months prior to Baseline
* History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator) within 3 months prior to Day 1
* An MS relapse that has occurred within the 50 days prior to randomization AND/OR the subject has not stabilized from a previous relapse prior to randomization
* Known history of, or positive screening test result for hepatitis C virus or hepatitis B virus
* Varicella or herpes zoster virus infection or any severe viral infection within 6 weeks before screening
* Exposure to varicella zoster virus within 21 days before screening

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1841 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (228):
- United States (46):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Naples, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Worchester, Massachusetts
  - Research Site, Clinton Township, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Latham, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
- Australia (6):
  - Research Site, Camperdown, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Woodville, South Australia
  - Research Site, Fitzroy, Victoria
  - Research Site, Heidelberg West, Victoria
- Brazil (8):
  - Research Site, Belo Horizonte, Estado de Bahia
  - Research Site, Brasília, Federal District
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande
  - Research Site, São Paulo, Rio Grande
  - Research Site, Campinas, São Paulo
  - Research Site, Ribeirão Preto, São Paulo
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Regina, Saskatchewan
- Czechia (10):
  - Research Site, Brno, Jihočeský kraj
  - Research Site, Jihlava, Kraj Vysočina
  - Research Site, Olomouc, Olomoucký kraj
  - Research Site, Prague, Prague
  - Research Site, Havířov, Severomoravksy Krav
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Ostrava
  - Research Site, Pardubice
- Denmark (4):
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Glostrup Municipality
  - Research Site, Odense C
- Finland (5):
  - Research Site, Oulu, Oulu
  - Research Site, Tampere, Western Finalnd
  - Research Site, Helsinki
  - Research Site, Seinäjoki
  - Research Site, Turku
- France (14):
  - Research Site, Strasbourg, Alsace
  - Research Site, Lyon, Auvergne-Rhône-Alpes
  - Research Site, Caen, Basse-normandie
  - Research Site, Amiens, Picardie
  - Research Site, Nice, Provence-Alpes-Côte d'Azur Region
  - Research Site, Bourdeaux
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lomme
  - Research Site, Marseille
  - Research Site, Nancy
  - Research Site, Toulouse
  - Research Site, Bobigny, Île-de-France Region
  - Research Site, Paris, Île-de-France Region
- Research Site, Tbilisi, Georgia
- Germany (15):
  - Research Site, Bad Mergentheim, Baden-Wurttemberg
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Bamberg, Bavaria
  - Research Site, Bayreuth, Bavaria
  - Research Site, München, Bavaria
  - Research Site, Neuburg an der Donau, Bavaria
  - Research Site, Hamburg, Hamburg
  - Research Site, Marburg, Hesse
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Trier, Rhineland-Palatinate
  - Research Site, Dresden, Saxony
  - Research Site, Berlin, State of Berlin
  - Research Site, Tübingen
- Greece (3):
  - Research Site, Athens, Attica
  - Research Site, Heraklion, Crete
  - Research Site, Thessaloniki, Macedoni
- Hungary (7):
  - Research Site, Budapest, Budapest
  - Research Site, Székesfehérvár, Fejér
  - Research Site, Győr, Győr-Moson-Sopron
  - Research Site, Esztergom
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Veszprém
- India (7):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Delhi, Dwivdee
  - Research Site, Bangalore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, New Delhi
- Research Site, Dublin, Dublin, Ireland
- Israel (7):
  - Research Site, Ashkelon, Ashqelon
  - Research Site, Tzrifin, Beer Yaakov
  - Research Site, Petah Tikva, Petah Tiqwa
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Tzfat
- Italy (10):
  - Research Site, Bari, Bari
  - Research Site, Cagliari, Cagliari
  - Research Site, Catania, Catania
  - Research Site, Genova, Genova
  - Research Site, Cefalù, PA
  - Research Site, Roma, Roma
  - Research Site, Orbassano, Torino
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
- Mexico (2):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
- Research Site, Chisinau, Moldova
- Poland (15):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Lublin, Lower Silesian Voivodeship
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Katowice, Silesian Voivodeship
  - Research Site, Kielce, Swietokrzycie
  - Research Site, Olsztyn, Warmian-Masurian Voivodeship
  - Research Site, Szczecin, West Pomeranian Voivodeship
  - Research Site, Bydgoszczas
  - Research Site, Plewiska
  - Research Site, Lódz, Łódź Voivodeship
- Romania (5):
  - Research Site, Bucurest, București
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Timișoara, Timiș County
  - Research Site, Iași
  - Research Site, Târgu Mures
- Russia (16):
  - Research Site, Kazan', Povolje-Tatarstan
  - Research Site, Yekaterinburg, Ural
  - Research Site, Yaroslavl, Yaroslavlr
  - Research Site, Chelyabinsk
  - Research Site, Kaluga
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Ufa
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Spain (6):
  - Research Site, Barcelona, Barcelona
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Córdoba, Cordoba
  - Research Site, Madrid, Madrid
  - Research Site, Seville, Sevilla
  - Research Site, Girona
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Malmo
  - Research Site, Stockholm
- Switzerland (2):
  - Research Site, Basel, Basel
  - Research Site, Lugano
- Ukraine (7):
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kyviv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Vinnitsa
  - Research Site, Zaporizhzhya
- United Kingdom (9):
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, New Castle Upon Tyne
  - Research Site, Nottingham
  - Research Site, Romford
  - Research Site, Salford
  - Research Site, Sheffield

REFERENCES:
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Castrogiovanni N, Mostert J, Repovic P, Bowen JD, Uitdehaag BMJ, Strijbis EMM, Cutter GR, Koch MW. Longitudinal Changes in Cognitive Test Scores in Patients With Relapsing-Remitting Multiple Sclerosis: An Analysis of the DECIDE Dataset. Neurology. 2023 Jul 4;101(1):e1-e11. doi: 10.1212/WNL.0000000000207301. Epub 2023 Apr 18. PMID 37072219
- [Derived] Cohan S, Kappos L, Giovannoni G, Wiendl H, Selmaj K, Havrdova EK, Rose J, Greenberg S, Phillips G, Ma W, Wang P, Lima G, Sabatella G. Efficacy of daclizumab beta versus intramuscular interferon beta-1a on disability progression across patient demographic and disease activity subgroups in DECIDE. Mult Scler. 2018 Dec;24(14):1883-1891. doi: 10.1177/1352458517735190. Epub 2017 Oct 6. PMID 28984179
- [Derived] Benedict RH, Cohan S, Lynch SG, Riester K, Wang P, Castro-Borrero W, Elkins J, Sabatella G. Improved cognitive outcomes in patients with relapsing-remitting multiple sclerosis treated with daclizumab beta: Results from the DECIDE study. Mult Scler. 2018 May;24(6):795-804. doi: 10.1177/1352458517707345. Epub 2017 May 9. PMID 28485186
- [Derived] Liu Y, Vollmer T, Havrdova E, Riester K, Lee A, Phillips G, Wang P, Sabatella G. Impact of daclizumab versus interferon beta-1a on patient-reported outcomes in relapsing-remitting multiple sclerosis. Mult Scler Relat Disord. 2017 Jan;11:18-24. doi: 10.1016/j.msard.2016.11.005. Epub 2016 Nov 13. PMID 28104250
- [Derived] Krueger JG, Kircik L, Hougeir F, Friedman A, You X, Lucas N, Greenberg SJ, Sweetser M, Castro-Borrero W, McCroskery P, Elkins J. Cutaneous Adverse Events in the Randomized, Double-Blind, Active-Comparator DECIDE Study of Daclizumab High-Yield Process Versus Intramuscular Interferon Beta-1a in Relapsing-Remitting Multiple Sclerosis. Adv Ther. 2016 Jul;33(7):1231-45. doi: 10.1007/s12325-016-0353-2. Epub 2016 Jun 1. PMID 27251051
- [Derived] Kappos L, Wiendl H, Selmaj K, Arnold DL, Havrdova E, Boyko A, Kaufman M, Rose J, Greenberg S, Sweetser M, Riester K, O'Neill G, Elkins J. Daclizumab HYP versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2015 Oct 8;373(15):1418-28. doi: 10.1056/NEJMoa1501481. PMID 26444729

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon Beta-1a: Interferon beta-1a (IFN β-1a) 30 µg intramuscular (IM) injection once weekly plus placebo to daclizumab high yield process (DAC HYP) subcutaneous (SC) once every 4 weeks for 96 to 144 weeks
- Daclizumab High Yield Process: DAC HYP 150 mg SC injection once every 4 weeks plus placebo to IFN β-1a intramuscular IM injection once weekly for 96 to 144 weeks
Period: Overall Study
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Started | 922 | 919
Completed | 694 | 724
Not Completed | 228 | 195
Not completed — Adverse Event | 47 | 56
Not completed — Lack of Efficacy | 46 | 23
Not completed — Lost to Follow-up | 12 | 9
Not completed — Consent Withdrawn | 98 | 80
Not completed — Investigator Decision | 4 | 6
Not completed — Death | 4 | 0
Not completed — Pregnancy | 4 | 7
Not completed — Noncompliance | 7 | 8
Not completed — Site Closure | 4 | 5
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Interferon Beta-1a: IFN β-1a 30 µg IM injection once weekly plus placebo to DAC HYP SC once every 4 weeks for 96 to 144 weeks
- Daclizumab High Yield Process: DAC HYP 150 mg SC injection once every 4 weeks plus placebo to IFN β-1a IM injection once weekly for 96 to 144 weeks
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process | Total
Number analyzed (Participants) | 922 | 919 | 1841
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.32) | 36.4 (9.36) | 36.3 (9.34)
Age, Customized [Number; unit: participants]
  18 to 19 years | 25 | 14 | 39
  20 to 29 years | 227 | 236 | 463
  30 to 39 years | 327 | 322 | 649
  40 to 49 years | 256 | 250 | 506
  50 to 55 years | 86 | 96 | 182
  > 55 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 627 | 625 | 1252
  Male | 295 | 294 | 589

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Annualized Relapse Rate (ARR)
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the examining neurologist. Only relapses confirmed by Independent Neurology Evaluation Committee (INEC) are included in this analysis. Adjusted ARR was estimated from a negative binomial regression model adjusted for the baseline relapse rate, history of prior IFN beta use, baseline Expanded Disability Status Scale score (EDSS; ≤ 2.5 vs > 2.5) and baseline age (≤ 35 vs > 35 years). Data after participants switched to alternative MS medications are excluded.
Time Frame: Up to 144 weeks
Population: participants with a relapse
Measure: Number (95% Confidence Interval); unit: relapses per person-years
Units Other Than Participants: Relapses
Groups:
- Daclizumab High Yield Process: DAC HYP 150 mg subcutaneous (SC) injection once every 4 weeks plus placebo to IFN β-1a intramuscular (IM) injection once weekly for 96 to 144 weeks
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Number analyzed (Participants) | 392 | 260
Number analyzed (Relapses) | 643 | 402
relapses per person-years | 0.393 [0.353 to 0.438] | 0.216 [0.191 to 0.244]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression — Estimated from a negative binomial regression model adjusted for the baseline relapse rate, history of prior IFN beta use, baseline EDSS (≤ 2.5 vs > 2.5) and baseline age (≤ 35 vs > 35 years); Rate Ratio = 0.550, 95% CI 2-sided [0.469 to 0.645]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; Percent Reduction = 45.0, 95% CI 2-sided [35.5 to 53.1]

2. Secondary Outcome: Adjusted Mean Number of New or Newly Enlarging T2 Hyperintense Lesions up to Week 96
Description: The quantity of lesions is assessed by brain magnetic resonance imaging (MRI). The adjusted mean number is estimated from a negative binomial regression model, adjusted for baseline volume of T2 from a negative binomial regression model, adjusted for baseline volume of T2 hyperintense lesions, history of prior IFN beta use and baseline age (≤ 35 vs > 35 years). To account for the timing of the MRI measurement, the logarithmic transformation of the scan number of the MRI assessment is included in the model as the 'offset' parameter. Observed data after participants switched to alternative MS medications are excluded. Missing data are not imputed. Only observed new or newly enlarging T2 lesions at the last visit of the participant up to Week 96 visit are used in this analysis.
Time Frame: up to 96 weeks
Population: participants with baseline and at least one post-baseline MRI measurement
Measure: Mean (95% Confidence Interval); unit: lesions
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Number analyzed (Participants) | 841 | 864
lesions | 9.44 [8.46 to 10.54] | 4.31 [3.85 to 4.81]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression — Estimated from a negative binomial regression model, adjusted for baseline volume of T2 hyperintense lesions, history of prior IFN beta use and baseline age (≤ 35 vs > 35 years); The logarithmic transformation of the scan number of the MRI assessment was included in the model as the 'offset' parameter; Percent Reduction = 54.4, 95% CI 2-sided [46.9 to 60.8]

3. Secondary Outcome: Proportion of Participants With Sustained Disability Progression at 144 Weeks
Description: Sustained disability progression is defined as: at least a 1.0-point increase on the EDSS from Baseline EDSS ≥ 1.0 that is sustained for 12 weeks, or at least a 1.5-point increase on the EDSS from baseline EDSS = 0 that is sustained for 12 weeks. The EDSS measures the disability status of people with MS on a scale that ranges from 0 to 10, with higher scores indicating more disability. Estimated proportion of participants with progression is based on the Kaplan-Meier product limit method. Participants were censored at the time of withdrawal/switch if they withdrew from study or switched to alternative MS medication without a progression. Participants with a tentative progression at the End of Treatment Period Visit (or the last EDSS assessment prior to alternative MS start date) and no confirmation assessment were censored at their last EDSS assessment.
Time Frame: Baseline through 144 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Number analyzed (Participants) | 922 | 919
proportion of participants | 0.203 | 0.162
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; p = 0.1575, Cox Proportional Hazard — Based on Cox Proportional Hazards model, adjusted by baseline EDSS values as continuous variable, history of prior IFN beta use, and baseline age (≤ 35 vs > 35 years); Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.66 to 1.07]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; Percent Reduction = 16.1, 95% CI 2-sided [-7.0 to 34.2]

4. Secondary Outcome: Proportion of Participants Relapse-free at Week 144
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the examining neurologist. Only relapses confirmed by INEC are included in this analysis. Data after participants switched to alternative MS medications are excluded. The estimated proportion of subjects relapse-free at Week 144 is based on the Kaplan-Meier product limit method.
Time Frame: 144 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Number analyzed (Participants) | 922 | 919
proportion of participants | 0.508 | 0.673
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard — Based on Cox proportional hazards model, adjusted for baseline relapse rate, history of prior IFN beta use, baseline EDSS (EDSS ≤ 2.5 vs EDSS > 2.5) and baseline age (≤ 35 vs > 35 years); Cox Proportional Hazard = 0.59, 95% CI 2-sided [0.50 to 0.69]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; Percent Reduction in Risk of Relapse = 40.9, 95% CI 2-sided [30.8 to 49.5]

5. Secondary Outcome: Percentage of Participants With a ≥ 7.5 Point Worsening From Baseline in the Multiple Sclerosis Impact Scale (MSIS-29) Physical Impact Score at 96 Weeks
Description: The MSIS-29 is a 29-item disease-specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures physical and psychological items. Worsening in the MSIS-29 physical score is defined as an increase of ≥ 7.5 points in the MSIS-29 physical score at 96 weeks compared to baseline. If a participant was missing data for less than 10 of the 20 items that make up the physical score, then the mean of the non-missing items were used for the missing items. If a participant was missing 10 or more of the 20 items that make up the physical score, or missing the questionnaire entirely, or if the questionnaire was completed after the participant switched to alternative MS medication, a random effects model was used to estimate the MSIS-29 physical score.
Time Frame: Baseline and 96 weeks
Population: participants with a baseline and Week 96 assessment
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta-1a | Daclizumab High Yield Process
Number analyzed (Participants) | 912 | 906
percentage of participants | 23 | 19
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; p = 0.0176, Regression, Logistic — Based on logistic regression model, adjusted for baseline MSIS-29 physical score, baseline Beck Depression Inventory (BDI) score, history of prior IFN beta use, and baseline age (≤ 35 vs > 35 years); Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.60 to 0.95]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Daclizumab High Yield Process; Test type: Superiority or Other; Percent Reduction in Odds of Worsening = 24.2, 95% CI 2-sided [4.7 to 39.6]

ADVERSE EVENTS:
Time Frame: All events were collected from Baseline through Week 164 (end of Post-dosing period).
Description: Treatment emergent events are reported. Events are considered treatment emergent if they occurred on or after the first dosing date and up to 180 days after the last dosing date.
Groups:
- IFN Beta-1a 30 mcg: IFN β-1a 30 µg IM injection once weekly plus placebo to DAC HYP SC once every 4 weeks for 96 to 144 weeks
- DAC HYP 150 mg: DAC HYP 150 mg subcutaneous (SC) injection once every 4 weeks plus placebo to IFN β-1a intramuscular (IM) injection once weekly for 96 to 144 weeks
Arm/Group | IFN Beta-1a 30 mcg | DAC HYP 150 mg
Serious Adverse Events (participants affected / at risk) | 194/922 | 221/919
Other Adverse Events (participants affected / at risk) | 783/922 | 731/919
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Beta-1a 30 mcg (N=922) | DAC HYP 150 mg (N=919)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 5
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Cystoid macular oedema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oroantral fistula (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Chronic tonsillitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 5
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Reiter's syndrome (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Strongyloidiasis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 8
Varicella (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 2
Viral myocarditis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 4
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 2
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Smear cervix abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Complex partial seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 4
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 3 | 2
Multiple sclerosis relapse (Nervous system disorders) | 124 | 97
Muscle spasticity (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Uhthoff's phenomenon (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 3
Depression suicidal (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Renal colic (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
Angioplasty (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 1
Ovarian cystectomy (Surgical and medical procedures) | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1
Spinal decompression (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Kawasaki's disease (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IFN Beta-1a 30 mcg (N=922) | DAC HYP 150 mg (N=919)
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 46
Diarrhoea (Gastrointestinal disorders) | 55 | 67
Nausea (Gastrointestinal disorders) | 46 | 46
Asthenia (General disorders) | 55 | 37
Fatigue (General disorders) | 76 | 69
Influenza like illness (General disorders) | 345 | 88
Injection site erythema (General disorders) | 47 | 40
Injection site pain (General disorders) | 102 | 96
Pyrexia (General disorders) | 134 | 104
Bronchitis (Infections and infestations) | 43 | 61
Influenza (Infections and infestations) | 56 | 82
Nasopharyngitis (Infections and infestations) | 197 | 226
Oral herpes (Infections and infestations) | 44 | 57
Pharyngitis (Infections and infestations) | 69 | 77
Upper respiratory tract infection (Infections and infestations) | 124 | 148
Urinary tract infection (Infections and infestations) | 96 | 92
Alanine aminotransferase increased (Investigations) | 66 | 69
Aspartate aminotransferase increased (Investigations) | 44 | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 | 71
Back pain (Musculoskeletal and connective tissue disorders) | 70 | 86
Myalgia (Musculoskeletal and connective tissue disorders) | 49 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 58 | 55
Dizziness (Nervous system disorders) | 37 | 48
Headache (Nervous system disorders) | 175 | 159
Hypoaesthesia (Nervous system disorders) | 54 | 54
Multiple sclerosis relapse (Nervous system disorders) | 428 | 293
Paraesthesia (Nervous system disorders) | 57 | 42
Depression (Psychiatric disorders) | 56 | 72
Insomnia (Psychiatric disorders) | 54 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 53
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 | 69
Rash (Skin and subcutaneous tissue disorders) | 26 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.